CLINICAL TRIAL: NCT00161447
Title: Male Hormonal Contraceptive Development: Suppression of Spermatogenesis With the Addition of a Potent Antagonist (Acyline) to Testosterone and DMPA (ACY-5)
Brief Title: Male Hormonal Contraceptive Development-ACY-5
Acronym: ACY-5
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); CONRAD (Other)
Responsible Party: William J Bremner, MD, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-0832-D; U54HD042454 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Contraception
Keywords: Male contraception; testosterone; acyline
MeSH Terms: interventions — acyline; Testosterone; Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Testosterone (T) gel for 6 months + DMPA (injected into muscle once)on Day 0 and at Month 3
  Interventions: Drug: Testosterone Gel; Drug: Depo-Medroxyprogesterone
- 2 (Active Comparator): Testosterone (T) gel for 6 months + DMPA (injected into muscle on Day 0 & at month 3) + Acyline (SQ) every two weeks for the first 12 weeks
  Interventions: Drug: Acyline; Drug: Testosterone Gel; Drug: Depo-Medroxyprogesterone

INTERVENTIONS:
Drug: Acyline — Acyline 300 mcg/kg SQ every 2 weeks for 12 weeks
  Arms: 2
Drug: Testosterone Gel — Testosterone Gel (10 g daily
  Other Names: Testim
Drug: Depo-Medroxyprogesterone — DMPA (injected into muscle) Day 0 & month 3
  Other Names: DMPA

SUMMARY:
The purpose of this research study is to help in the development of male contraception (birth control).

DETAILED DESCRIPTION:
The objective is to conduct a male contraceptive trial in which we will evaluate the suppressive effects of acyline when administered in combination with Testosterone (T) and the progestin depo-medroxyprogesterone acetate (DMPA).

We will be administering combinations of three drugs: Testosterone (T) by gel, Depot Medroxyprogesterone acetate (DMPA) and Acyline to see their effects on sperm production. The T/DMPA/Acyline combination will allow us to determine if the more rapid and complete gonadotropin suppression mediated by the early addition of a GnRH antagonist will accelerate and enhance suppression of spermatogenesis.

In prior studies with testosterone and DMPA these drug, which are hormones, have been found to be safe, and to reversibly suppress sperm counts to zero in about 80% of men. We hope to improve this to 100% of men by adding another drug, Acyline.

Acyline is an GnRH antagonist which blocks the release of LH and FSH from the pituitary. DMPA is approved by the FDA for use as a female contraceptive. The endpoint will be suppression of spermatogenesis to zero (azoospermia) by the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-55
* In good general health
* With normal sperm counts
* Willing to use an acceptable form of contraception

Exclusion Criteria:

* Men in poor health
* Significant chronic or acute medical illness
* Skin conditions that might interfere with or be exacerbated by testosterone gel
* Known history of alcohol, illicit drug or anabolic steroid abuse
* Abnormal reproductive function
* Participation in a long-term male contraceptive study within past three months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2004-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary biological end points in this trial will be suppression of spermatogenesis and gonadotropins while monitoring for any adverse changes in lipid metabolism, sexual side effects or in general health | One year

SECONDARY OUTCOMES:
Regimen acceptability, sexual function, glucose tolerance, intratesticular hormone levels | One year

CONTACTS AND LOCATIONS:
Overall Officials: William J Bremner, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Meriggiola MC, Bremner WJ, Costantino A, Di Cintio G, Flamigni C. Low dose of cyproterone acetate and testosterone enanthate for contraception in men. Hum Reprod. 1998 May;13(5):1225-9. doi: 10.1093/humrep/13.5.1225. PMID 9647551
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Kamischke A, Venherm S, Ploger D, von Eckardstein S, Nieschlag E. Intramuscular testosterone undecanoate and norethisterone enanthate in a clinical trial for male contraception. J Clin Endocrinol Metab. 2001 Jan;86(1):303-9. doi: 10.1210/jcem.86.1.7057. PMID 11232016
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Result] Page ST, Amory JK, Anawalt BD, Irwig MS, Brockenbrough AT, Matsumoto AM, Bremner WJ. Testosterone gel combined with depomedroxyprogesterone acetate is an effective male hormonal contraceptive regimen and is not enhanced by the addition of a GnRH antagonist. J Clin Endocrinol Metab. 2006 Nov;91(11):4374-80. doi: 10.1210/jc.2006-1411. Epub 2006 Aug 29. PMID 16940442
- [Result] Amory JK, Page ST, Anawalt BD, Matsumoto AM, Bremner WJ. Acceptability of a combination testosterone gel and depomedroxyprogesterone acetate male contraceptive regimen. Contraception. 2007 Mar;75(3):218-23. doi: 10.1016/j.contraception.2006.11.003. Epub 2007 Jan 16. PMID 17303493
- [Result] Page ST, Kalhorn TF, Bremner WJ, Anawalt BD, Matsumoto AM, Amory JK. Intratesticular androgens and spermatogenesis during severe gonadotropin suppression induced by male hormonal contraceptive treatment. J Androl. 2007 Sep-Oct;28(5):734-41. doi: 10.2164/jandrol.107.002790. Epub 2007 May 9. PMID 17494097